CLINICAL TRIAL: NCT00745394
Title: Validation of Somatic and Cerebral Near Infrared Spectroscopy (NIRS) During Cardiopulmonary Bypass In Pediatric Patients: A Prospective Clinical Study
Brief Title: Validation of Near Infrared Spectroscopy (NIRS) During Heart-Lung Bypass in Children
Acronym: NIRS
Status: Withdrawn | Type: Observational
Why Stopped: No patient has been enrolled in this study for more than 8 years. Study closed.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Sponsor
Other Study IDs: 072007-057
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Bypass
Keywords: NIRS; bypass; cardiopulmonary; CPB; monitoring; system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-invasive assessment of blood flow to organs has long challenged clinicians. Recently, near infrared spectroscopy (NIRS) has been recognized as a methodology that may achieve this goal. A commercially available NIRS monitor, marketed by Somanetics, Inc., is now in widespread use in the clinical care of pediatric cardiac patients in the operating room and in the intensive care unit post-operatively. When a patch/probe from the monitor is placed on the forehead or lower back, blood oxygen concentration data is obtained which has been found to correlate with actual blood samples taken by IV. The presence of this NIRS data would give the surgeon important feedback about blood flow to important areas like the brain and kidneys during heart surgeries on children and after the operation is completed in the intensive care unit.

The investigator wishes to perform a prospective study of the NIRS monitor use with children that need heart surgeries that require heart-lung bypass and sometimes require monitoring in the ICU, post-operatively.

DETAILED DESCRIPTION:
After patients are prospectively consented pre-operatively, standard medical care, including the use of the NIRS monitor, will be implemented during the patient's operation and post-operatively in the intensive care unit with few modifications. These modifications include: (1) the placement of an oximetric probe in the lumen of the cardiopulmonary bypass circuit tubing which will output continuous blood oxygen content during bypass, (2) the addition of extra connectors to the bypass tubing to allow blood draws during surgery, (3) placement of doppler blood flow probes on the tubing to measure blood flow velocity, and (4) the addition of LFTs during the post-operative phase, if followed. Patients that receive operations that require circulatory arrest and/or selective cerebral perfusion will be followed in the ICU for 5 days. Data from the bypass machine along, data collected from the NIRS and oximetric probe monitor, and serum data will be interfaced into a data collection system.

Data to be collected: Minimum patient demographic data (age, sex, ethnic origin), NIRS data, serum blood gas data, serum lactate levels, hemoglobin levels, vital signs, doppler blood flow data, LFT analysis, clinical course events/data (i.e. need for dialysis, length of stay, surgical time points, etc), diagnostic test results (EKGs, ECHOs, etc), significant medical history data, and standard of care laboratory results.

The investigator wishes to evaluate the relationship of this data with the patient's diagnosis, operation performed, post-operative course, and outcome. Validation of the use of the NIRS monitor and further characterization of the NIRS monitor will also be sought.

Notes: 1/15/2025 -Record transferred from Ann & Robert H Lurie Children's Hospital of Chicago to University of Texas Southwestern Medical Center since Record shows UTSW as the Sponsor. Dr. Forbess (Responsible Party) and his team for this study no longer at UTSW to shed light on why this record was transferred to Lurie Children's in 2019. Dr. Jaquiss from Cardiovascular & Thoracic Surgery Department at UTSW confirmed on 1/7/2025 that - "No patient has been enrolled in this study and should be considered to be closed".

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients that require cardiopulmonary bypass during surgical correction of heart disease
* 2. Prospective, Informed Consent

Exclusion Criteria:

* 1. Patients with malformations of venous return to the heart (e.g. interrupted IVC with azygous continuation).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who undergo surgical correction of their congenital heart disease that require cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Determine correlation between cerebral/somatic NIRS saturation data obtained on CPB and oxygen saturation and lactate data obtained from the superior vena caval (SVC) blood. | Length of surgery with possible 5 day follow-up in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Forbess, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Medical Center, Dallas, Texas, United States